CLINICAL TRIAL: NCT04366778
Title: Evaluation of TEM-tPA (Thromboelastometry With tPA) to Detect Covid-19 Patients at High Risk of Thrombosis
Brief Title: Thrombosis and Covid-19
Acronym: COVBIO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0401 - COVBIO; ID-RCB (Other: 2020-A01193-36)
Record Dates: First submitted 2020-04-23; First posted 2020-04-29 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Thrombosis; Covid-19; SARS-CoV 2
MeSH Terms: conditions — Thrombosis; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients hospitalized for Covid-19: Patients with Covid-19 infection hospitalized in Lyon University Hospitals
  Interventions: Diagnostic Test: TEM-tPA
- patients hospitalized for Covid-19 who present thrombosis: Patients with Covid-19 infection hospitalized in Lyon University Hospitals who present thrombosis during hospitalization
  Interventions: Diagnostic Test: TEM-tPA

INTERVENTIONS:
Diagnostic Test: TEM-tPA — 325 patients with Covid-19 hospitalized in Lyon University Hospitals will have TEM-tPA measurements in parallel to D-dimers every 3 days during the hospitalization period. TEM-tPA of patients with and without thrombosis will be compared and their fibrinolysis (PAI-1, TAFI, tPA, thrombin) will be further explored.

SUMMARY:
The coronavirus disease of 2019 (COVID-19) is a viral illness caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV2), now deemed a pandemic by the World Health Organization. Some COVID-19 patients may develop coagulopathy which is associated with poor prognosis and high risk of thrombosis. Some patients develop severe thrombotic complications, such as pulmonary embolism, despite anti-thrombotic prophylaxis by low molecular weight heparin. The aim of this project is to evaluate modified thromboelastometry for identifying patients at high risk of thrombosis. The hypothesize is that hypofibrinolysis with increased plasma PAI-1, TAFI (thrombin-activatable fibrinolysis inhibitor ) levels in association with high thrombin generation may explain high incidence of thrombosis in this population. A simple laboratory assay, widely available in hospitals, such as thromboelastometry, might be of great clinical interest to detect Covid-19 patients with high risk of thrombosis. In order to make ROTEM more sensitive to hypofibrinolysis, exogenous t-PA will be added in the assay. The preliminary results showed that patients with Covid-19 have significant hypercoagulability detectable with ROTEM and Covid-19 patients with thrombosis have both hypercoagulability and hypofibrinolysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Covid-19
* non-opposition of the patient to participate

Exclusion Criteria:

* Non-Covid-19 acute respiratory distress syndrome
* Non-Covid septicemia
* Pregnant women
* Breastfeeding women
* Protected vulnerable adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed diagnosis of Covid-19 (PCR test positive or clinical signs associated with lung CR scan showing typical Covid-19 manifestation)
Sampling Method: Non-Probability Sample
Enrollment: 341 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Coagulability | Day 0
  TEM-tPA profile of patients will be defined with a combination of the following parameters :
  Maximal Clot Firmness (MCF) (mm) alpha angle (°) Lysis Index (LI) 30 (%) Lysis Onset Time (LOT) (min)
Coagulability | Day 3
  TEM-tPA profile of patients will be defined with a combination of the following parameters :
  Maximal Clot Firmness (MCF) (mm) alpha angle (°) Lysis Index (LI) 30 (%) Lysis Onset Time (LOT) (min)
Coagulability | Day 6
  TEM-tPA profile of patients will be defined with a combination of the following parameters :
  Maximal Clot Firmness (MCF) (mm) alpha angle (°) Lysis Index (LI) 30 (%) Lysis Onset Time (LOT) (min)
Coagulability | Day 9
  TEM-tPA profile of patients will be defined with a combination of the following parameters :
  Maximal Clot Firmness (MCF) (mm) alpha angle (°) Lysis Index (LI) 30 (%) Lysis Onset Time (LOT) (min)
Coagulability | Day 12
  TEM-tPA profile of patients will be defined with a combination of the following parameters :
  Maximal Clot Firmness (MCF) (mm) alpha angle (°) Lysis Index (LI) 30 (%) Lysis Onset Time (LOT) (min)
Coagulability | Day 15
  TEM-tPA profile of patients will be defined with a combination of the following parameters :
  Maximal Clot Firmness (MCF) (mm) alpha angle (°) Lysis Index (LI) 30 (%) Lysis Onset Time (LOT) (min)
Venous thrombotic event (VTE) or arterial thrombosis | Day 15
  Occurence of VTE or arterial thrombosis during hospitalization :
  * Pulmonary embolism diagnosed with CT scan
  * Venous or arterial thrombosis diagnosed with ultrasound exam

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Louis Pradel, Bron, France

IPD SHARING:
Plan to Share IPD: No